CLINICAL TRIAL: NCT06854406
Title: Varenicline in the Treatment of Visceral Sensation: A Pilot Study
Brief Title: A Study of Varenicline in the Treatment of Visceral Sensation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-013815
Record Dates: First submitted 2025-02-21; First posted 2025-03-03 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; pain
MeSH Terms: conditions — Irritable Bowel Syndrome; Pain | interventions — Varenicline

STUDY DESIGN:
Intervention Model Description: To evaluate the effect of varenicline on rectal sensation, based on ascending method of limits and on graded rapid phasic distensions in participants with non-constipation IBS and chronic abdominal pain
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Varenicicline (Experimental): Varenicline is a α4β2 and α6β2 partial agonist.
  Varenicline (Chantix) is an FDA-approved partial agonist at α4β2 and α6β2 nAChRs with documented efficacy in the management of chronic pain associated with opioid withdrawal
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Initial, 0.5 mg orally once daily for 3 days, then 0.5 mg every 12 hours on days 4 through 7, and then 1 mg in morning of day 8. Medication is taken after eating and with a full glass of water.

SUMMARY:
The purpose of this study is to evaluate the effect of varenicline on rectal sensation, based on ascending method of limits and on graded rapid phasic distensions in participants with non-constipation IBS and chronic abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be 18-70 years of age
2. Irritable bowel syndrome with pain, but no constipation [that is IBS-D (diarrhea), IBS-M (mixed), or IBS-U (unspecified)]

Exclusion Criteria:

1. Diagnosis of moderate-severe depression as per HADS>8
2. Alcohol or illicit substance dependence or abuse in the past 12 months
3. Dementia, unprovoked seizure history, seizure disorder
4. Pregnancy (all women of childbearing potential will be required to have a negative pregnancy test prior to initiation, and will be on a highly effective method of contraception, as detailed in the consent form)
5. Significant change or increase in antidepressant or pain medications within the last four weeks; significant change in primary treatment interventions for pain in the past four weeks
6. Medically unstable
7. Severe hepatic or renal impairment, such as baseline AST or ALT >2.5 X upper normal limit or end-stage renal disease with estimated glomerular filtration rate or creatinine clearance <15 mL/min
8. Concomitant use of strong CYP3A4 inhibitors and strong or moderate CYP3A4 inducers

Note: Other protocol defined Inclusion/Exclusion Criteria may apply.

Eligibility last updated 12/27/2024. Questions regarding updates should be directed to the study team contact.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Rectal compliance | Comparison on day 8 of vareniciline treatment compared to baseline
  Pressure-volume relationship of rectum during balloon distension
Rectal sensation thresholds during ascending method of limits | Comparison on day 8 of vareniciline treatment compared to baseline
  Report of rectal sensation during balloon distension 0-44mmHg
Rectal sensation ratings during random order, graded phasic distensions | Comparison on day 8 of vareniciline treatment compared to baseline
  Report of rectal sensation during balloon distensions

SECONDARY OUTCOMES:
Safety/adverse effects | 8 days
  Safety/adverse effects during administration of varenicicline

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No